CLINICAL TRIAL: NCT02219659
Title: Comparing Strategies of Pairing Sedation and Weaning Protocols on Outcomes of Mechanical Ventilation: A Pilot Study
Brief Title: Pilot Study on Pairing Sedation Strategies and Weaning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Collaborators: Memorial Medical Center Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25613
Record Dates: First submitted 2014-02-20; First posted 2014-08-19 (Estimated); Results first posted 2024-05-14 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Failure
Keywords: sedation strategy; mechanical ventilation; ventilator weaning
MeSH Terms: interventions — Fentanyl; Midazolam; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sedation protocol with interruption (Active Comparator): Continuous infusion of fentanyl and midazolam is started per protocol. Both drugs are titrated to target pain score (0 to 3) using Critical Care Pain Observation Tool (CPOT) and target sedation score (0 to -3) using Richmond Agitation Sedation Scale (RASS). Every morning both drugs are stopped (Daily Interruption) and patient's wakefulness is assessed per protocol. If patient's pain and RASS score stays within the target, both drugs are kept off. If patient shows any signs and symptoms of pain or agitation (described in the study protocol), both drugs are restarted at a half dose of the previous dose and titrated to target pain and RASS score. Every morning both drugs are stopped and when patient is awake and met the SBT safety screen, 120-min continuous positive airway pressure (CPAP) trial is performed.
  Interventions: Drug: Sedation Protocol with Daily Interruption
- Sedation protocol without Interruption (Active Comparator): Continuous infusion of fentanyl and midazolam is started per protocol. Both drugs are titrated to target pain score (0 to 3) using Critical Care Pain Observation Tool (CPOT) and target sedation score (0 to -3) using Richmond Agitation Sedation Scale (RASS). Daily interruption of fentanyl and midazolam is not performed. Every morning 120-min CPAP trial is performed as long as the patient's RASS score is 0 to -2 and the patient passes the SBT safety screen.
  Interventions: Drug: Sedation Protocol Without Daily Interruption
- Fentanyl push first (Active Comparator): This arm attempts to manage patient's pain and agitation with analgesia first. Fentanyl intravenous (IV) pushes are administered every 5 minutes as needed to target pain and sedation score, up to 4 doses per hour. Every morning 120-min CPAP trial is performed as long as patient's RASS score is 0 to -2 and patient passes the SBT safety screen. If fentanyl IV push doses alone cannot manage patient's pain and agitation (could not reach the target score), notify the study team. Fentanyl infusion is started and titrated to target pain and sedation score up to 6 hours. If fentanyl infusion is titrated up twice consecutively and target pain and sedation score are not met, notify the study team. Propofol infusion is started and titrated to target RASS score up to 6 hours.
  Interventions: Drug: Fentanyl Push First

INTERVENTIONS:
Drug: Sedation Protocol with Daily Interruption — Continuous infusion of fentanyl and midazolam is started and titrated to target pain and RASS score: Fentanyl started at 25 mcg/hr titrated by 25 mcg/hr every 30 minutes to goal pain score; Midazolam started at 1 mg/hr titrated by 1 mg/hr every hour to goal RASS score for the study design duration (28 days) or for the duration of mechanical ventilation. Every morning both infusions are stopped and when the patient is awake and met the SBT safety screen, 120-min CPAP trial is performed. If the patient meets the CPAP passing criteria, arterial blood gas (ABG) is done and the patient is placed back to the previous ventilator setting. ABG result is notified to the physician for determination for extubation. If the patient does not pass the CPAP trial it is repeated next morning.
  Other Names: fentanyl; midazolam
  Arms: Sedation protocol with interruption
Drug: Sedation Protocol Without Daily Interruption — Continuous infusion of fentanyl and midazolam is started and titrated to target pain and RASS score: Fentanyl started at 25 mcg/hr titrated by 25 mcg/hr every 30 minutes to goal pain score; Midazolam started at 1 mg/hr titrated by 1 mg/hr every hour to goal RASS score for the study design duration (28 days) or for the duration of mechanical ventilation. Every morning when the patient's RASS score is 0 to -2 and the patient passes the SBT safety screen, 120-min CPAP trial is performed. If the patient meets the CPAP passing criteria, arterial blood gas (ABG) is done and the patient is placed back to the previous ventilator setting. ABG result is notified to the physician for determination for extubation. If the patient does not pass the CPAP trial it is repeated next morning.
  Other Names: fentanyl; midazolam
  Arms: Sedation protocol without Interruption
Drug: Fentanyl Push First — Fentanyl 25 mcg intravenous push (IVP) every 5 min up to 4 doses hourly as needed to target pain score for the study design duration (28 days) or for the duration of mechanical ventilation. Every morning when patient's RASS is 0 to -2 and passes the SBT safety screen, 120-min CPAP trial is performed. If patient meets CPAP passing criteria, the physician will be notified for determination of extubation. If patient does not pass, it is repeated next morning. If target RASS is not achieved with fentanyl IV push alone, study team is notified and fentanyl infusion at 50 mcg/hr titrated by 25 mcg/hr every 30 min to target pain score (max 6 hrs). If target RASS score is not achieved with the fentanyl IV, propofol infusion is started at 5 mcg/kg/hr titrated by 5 mcg/kg/hr every 15 min to target RASS score (max 6 hrs).
  Other Names: fentanyl; propofol
  Arms: Fentanyl push first

SUMMARY:
A three-arm, randomized, pilot study, to assess the feasibility for the analgesia-first sedation (AFS) study arm/intervention (Fentanyl push first). The study will assess additional outcomes for all three (3) validated strategies for sedation and pain management.

DETAILED DESCRIPTION:
A three-arm, randomized, pilot study, to assess the feasibility for the analgesia-first sedation (AFS) study arm/intervention (Fentanyl push first). The study will assess additional outcomes for all three (3) validated strategies for sedation and pain management.

A significant proportion of patients admitted to the intensive care unit (ICU) require mechanical ventilation (MV). To maintain comfort and facilitate quality care, large quantities of sedatives and analgesics are often administered either by continuous infusion, with or without daily interruption (DI) of sedation, or as intermittent doses of analgesics. Three validated sedation strategies are currently available. A recently published study ( trial has shown that instituting protocol-directed sedation in patients requiring continuous infusion of sedatives and analgesics, whether or not daily interruption (DI) of the sedative occurs, will improve MV outcomes, specifically the duration of MV. Girard et al performed a randomized, multicenter, clinical trial (ABC- Awakening and Breathing Controlled trial) evaluating the pairing of a spontaneous awakening trial (SAT) with an SBT. Most recently, a Danish study by Strom et al. investigated whether an analgesia-first approach to patient comfort that consisted of intermittent doses of intravenous opioids, and the initiation of IV sedation for short periods only when acute agitation was present, would be superior to a protocol similar to the ABC trial. While the three above mentioned approaches are accepted and currently implemented in the critical care community there is no comparative study or evaluation on the optimal timing to conduct a spontaneous breathing trial (SBT) for assessing weaning readiness with each of these strategies. It is possible that a SAT strategy, where sedative and opioid infusions are interrupted, may lead to more agitation and anxiety than a strategy in patients managed with a sedation protocol where intravenous sedative and analgesic therapy is regularly titrated to maintain patients in a lightly sedated state. Moreover, it remains unclear whether analgesia-first strategy (AFS) is feasible and if there are advantages of AFS (Fentanyl push first interventions) over either an SAT or sedation protocol strategy in terms of the time it takes to wean patients from MV or ICU length of stay. However, it is noteworthy to mention that the analgesia-first strategy was associated with more delirium episodes, which were attributed to the ability to assess for it in a more awake patient. However, comparing delirium occurrence in studies with different sedation goals and methodologies may be inaccurate.

The investigators therefore propose a three-arm, randomized clinical trial. This pilot study will measure feasibility for the implementation of analgesia-first sedation (AFS) study arm/intervention (Fentanyl push first). The study will assess additional outcomes for all three (3) validated strategies for sedation and pain management.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Mechanically ventilated with an expected duration of MV ≥ 48 hours
3. ICU team has initiated continuous sedative and/or /analgesic infusions

Exclusion criteria:

1. Admission after resuscitation from cardiac arrest
2. Admission with traumatic brain injury or another acute neurologic event (e,g. stroke, uncontrolled seizures).
3. History of severe dementia
4. Admission because of acute alcohol withdrawal or acute drug intoxication
5. Administration of more than 24 hours of continuous sedation
6. Allergy to fentanyl, midazolam, and/or propofol
7. Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-12; Primary Completion 2017-05 (Actual); Study Completion 2018-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maged Tanios, MD, MPH, Principal Investigator — Long Beach Memorial Medical Center
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12-2014 to 5/2017, ICU
Groups:
- Fentanyl Push First: Fentanyl intravenous (IV) pushes are administered every 5 minutes as needed to target pain and sedation score, up to 4 doses per hour. If fentanyl IV push doses alone cannot manage patient's pain and agitation (could not reach the target score), notify the study team. Fentanyl infusion is started and titrated to target pain and sedation score up to 6 hours. If fentanyl infusion is titrated up twice consecutively and target pain and sedation score are not met, notify the study team. Propofol infusion is started and titrated to target RASS score up to 6 hours.
  Fentanyl Push First: Fentanyl 25 mcg intravenous push (IVP) every 5 min up to 4 doses hourly as needed to target pain score for the study design duration (28 days) or for the duration of mechanical ventilation. Every morn
- Sedation Protocol Without Interruption: Continuous infusion of fentanyl and midazolam is started per protocol. Both drugs are titrated to target pain score (0 to 3) using Critical Care Pain Observation Tool (CPOT) and target sedation score (0 to -3) using Richmond Agitation Sedation Scale (RASS). Daily interruption of fentanyl and midazolam is not performed. Every morning 120-min CPAP trial is performed as long as the patient's RASS score is 0 to -2 and the patient passes the SBT safety screen.
  Sedation Protocol Without Daily Interruption: Continuous infusion of fentanyl and midazolam is started and titrated to target pain and RASS score: Fentanyl started at 25 mcg/hr titrated by 25 mcg/hr every 30 minutes to goal pain score; Midazolam started at 1 mg/hr titrated by 1 mg/hr every hour to goal RASS score for the study design duration (28 days) or for the duration of mechanical ventilation. Every morning when the patient's RASS score is 0 to -2 and the patient passes the SBT safety screen, 120-min CPAP trial is performed.
Period: Overall Study
Arm/Group | Fentanyl Push First | Sedation Protocol Without Interruption | Sedation Protocol With Interruption
Started | 29 | 30 | 31
Completed | 27 | 28 | 31
Not Completed | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fentanyl Push First: . Fentanyl intravenous (IV) pushes are administered every 5 minutes as needed to target pain and sedation score, up to 4 doses per hour. Every morning 120-min CPAP trial is performed as long as patient's RASS score is 0 to -2 and patient passes the SBT safety screen. If fentanyl IV push doses alone cannot manage patient's pain and agitation (could not reach the target score), notify the study team. Fentanyl infusion is started and titrated to target pain and sedation score up to 6 hours. If fentanyl infusion is titrated up twice consecutively and target pain and sedation score are not met, notify the study team. Propofol infusion is started and titrated to target RASS score up to 6 hours.
- Total: Total of all reporting groups
Arm/Group | Fentanyl Push First | Sedation Protocol Without Interruption | Sedation Protocol With Interruption | Total
Number analyzed (Participants) | 27 | 28 | 31 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 13 | 15 | 40
  >=65 years | 15 | 15 | 16 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (15.8) | 64.1 (18.4) | 66 (16.4) | 65.2 (18.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 8 | 10
  Male | 26 | 27 | 23 | 76
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 28 | 31 | 86
Body Mass Index (BMI) Kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) Kg/m^2
  kg/m^2 | 31.5 (9.9) | 31.2 (10.1) | 30.3 (10.3) | 31 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility
Description: Study feasibility for all 3 Arms/Groups (i.e., "Fentanyl Push First", "Sedation Protocol Without Interruption", and "Sedation Protocol with Interruption") being greater than or equal to 80% and protocol feasibility was based on protocol compliance (total percentage of study days participants were compliant with protocol).
Time Frame: Up to 28 days
Population: All 3 arms were measure, and the measurement was based on total % of study days where compliant with the respective protocol.
Measure: Number; unit: Percentage of study days
Groups:
- Protocol Compliance: Feasibility outcomes and a priori-deﬁned benchmarks: protocol compliance
- Sedation Protocol With Interruption: Continuous infusion of fentanyl and midazolam is started per protocol. Both drugs are titrated to target pain score (0 to 3) using Critical Care Pain Observation Tool (CPOT) and target sedation score (0 to -3) using Richmond Agitation Sedation Scale (RASS). Every morning both drugs are stopped (Daily Interruption) and patient's wakefulness is assessed per protocol. If patient's pain and RASS score stays within the target, both drugs are kept off. If patient shows any signs and symptoms of pain or agitation (described in the study protocol), both drugs are restarted at a half dose of the previous dose and titrated to target pain and RASS score. Every morning both drugs are stopped and when patient is awake and
Arm/Group | Protocol Compliance | Sedation Protocol Without Interruption | Sedation Protocol With Interruption
Number analyzed (Participants) | 27 | 28 | 31
Percentage of study days | 91 | 97 | 93

2. Secondary Outcome: ICU Length of Stay
Description: Duration of ICU stay at 28 days
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fentanyl Push First | Sedation Protocol Without Interruption | Sedation Protocol With Interruption
Number analyzed (Participants) | 27 | 28 | 31
Days | 7 [4 to 14] | 7 [3 to 15] | 8 [3 to 15]

3. Other Pre Specified Outcome: Mechanical Ventilation Free Days
Description: This is clinical outcome and represent the number of days where patients were breathing without assistance during the study period.
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fentanyl Push First | Sedation Protocol Without Interruption | Sedation Protocol With Interruption
Number analyzed (Participants) | 27 | 28 | 31
days | 24 [23 to 26] | 23.5 [20 to 26] | 24 [21 to 26]

4. Other Pre Specified Outcome: Duration of Weaning
Description: Duration of weaning: Time from initiation of weaning until successful extubation
Time Frame: Up to 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fentanyl Push First | Sedation Protocol Without Interruption | Sedation Protocol With Interruption
Number analyzed (Participants) | 27 | 28 | 31
days | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: 28 days
Description: Unintentional extubation
Arm/Group | Fentanyl Push First | Sedation Protocol Without Interruption | Sedation Protocol With Interruption
All-Cause Mortality (participants affected / at risk) | 8/27 | 6/28 | 4/31
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/28 | 1/31
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28 | 0/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Push First (N=27) | Sedation Protocol Without Interruption (N=28) | Sedation Protocol With Interruption (N=31)
Unplanned Extubation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 — Unplanned extubation (UE) is the unintentional and uncontrolled removal of an endotracheal tube (ETT).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT02219659/Prot_SAP_000.pdf